CLINICAL TRIAL: NCT01767298
Title: Pharmacokinetic Interactions of Valsartan and Hydrochlorothiazide: An Open-Label, Randomized, Four-Period Crossover Study in Healthy Egyptian Male Volunteers (PART II)
Brief Title: Pharmacokinetic Interactions of Valsartan and Hydrochlorothiazide (Double Doses)
Acronym: PKVH PART II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Sally Helmy, PhD, CPHQ, Lecturer of Pharmaceutics, Faculty of Pharmacy, Damanhour University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PPT1 PART II
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Normotensive Participants
Keywords: Fixed dose combination; Pharmacokinetics; Valsartan; Hydrochlorothiazide
MeSH Terms: interventions — Valsartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Valsartan 320 mg alone (Other): Valsartan alone
  Interventions: Drug: Valsartan
- Hydrochlorothiazide 25 mg alone (Other): Hydrochlorothiazide alone
  Interventions: Drug: Hydrochlorothiazide
- Valsartan 320 mg + Hydrochlorothiazide 25 mg (Other): Concomitant administration of valsartan 320 mg + Hydrochlorothiazide 25 mg
  Interventions: Drug: Valsartan/Hydrochlorothiazide
- Valsartan / Hydrochlorothiazide 320 mg/25mg (Other): Fixed dose combination of valsartan 320 mg + Hydrochlorothiazide 25 mg
  Interventions: Drug: Valsartan/Hydrochlorothiazide

INTERVENTIONS:
Drug: Valsartan/Hydrochlorothiazide — Co-administration or fixed dose combination
  Arms: Valsartan / Hydrochlorothiazide 320 mg/25mg; Valsartan 320 mg + Hydrochlorothiazide 25 mg
Drug: Valsartan — Valsartan alone
  Arms: Valsartan 320 mg alone
Drug: Hydrochlorothiazide — Hydrochlorothiazide alone
  Arms: Hydrochlorothiazide 25 mg alone

SUMMARY:
This study was conducted to compare the rate and extent of absorption of valsartan and hydrochlorothiazide. To maximize the possibility of finding drug-drug interactions, the dose of valsartan and hydrochlorothiazide was doubled (320 mg of VAL and 25 mg of HCT).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and not more than 45 healthy male volunteers
* Actual weight no more than ± 30% from ideal body weight based on sex, height, and body frame
* Who had passed all the screening parameters
* Free of any drug exposure known to interfere with the pharmacokinetics or assay of fexofenadine for at least 10 days prior to the study
* Who had to be able to communicate effectively with study personnel, be literate, and able to give consent.

Exclusion Criteria:

* A clinically significant abnormal physical exam, medical history, or laboratory studies
* If they showed a sitting SBP of >140 or <100 mmHg, DBP > 90 or <60mm Hg, or a pulse rate of > 95 or < 50 beats/min at screening
* A history of serious intolerance, allergy, or sensitivity to fexofenadine
* The use of any prescription drug within the previous month or use of any over-the-counter medication (with the exception of acetaminophen) within the past 14 days
* A history of blood dyscrasias
* A history of alcohol or drug abuse within the past year
* Donation of blood during the 8 weeks prior to the study or plans to donate blood during or within 8 weeks of completing the study
* Unable to tolerate vein puncture and multiple blood samplings
* Any surgical/medical condition that might alter drug absorption, distribution, metabolism, or excretion
* Cannot follow instructions, in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Tolerability | Participants will be followed for the duration of study, an expected average of 6 weeks.
  Tolerability was assessed based on changes in vital signs (temperature, blood pressure, pulse, and heart rate), measured before dosing in each period and approximately every 4 hours thereafter, and laboratory tests (hematology, biochemistry, liver function, and urinalysis), and performed at baseline and at the end of the study. In addition, a physician questioned volunteers about any adverse events occurring during the study, addressed them as necessary, and recorded them on the appropriate form. This physician was not blinded to treatment, but had no involvement in the study.